CLINICAL TRIAL: NCT04997421
Title: Safety and Efficacy of HA380 HEMoadsorption in Combination With OXiris Membrane for Continuous HemoDiaFiltration in Patients With Septic Shock - HEMOX-HDF Trial
Brief Title: Safety and Efficacy of HA380 Hemoadsorption in Patients With Septic Shock
Acronym: HEMOX-HDF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T96/2021
Record Dates: First submitted 2021-06-21; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVVHDF with Oxiris®-AN69 membrane (Active Comparator): Control arm
  Interventions: Device: Continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes
- CVVHDF with Oxiris®-AN69 membrane + Hemoadsorption using HA380 (Active Comparator): Intervention arm
  Interventions: Device: Combined HA380 hemoadsorption and continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes

INTERVENTIONS:
Device: Combined HA380 hemoadsorption and continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes — Combined HA380 hemoadsorption and continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes (intervention arm)or mere CVVHDF using the Oxiris®-AN69 membrane (control arm).
  Arms: CVVHDF with Oxiris®-AN69 membrane + Hemoadsorption using HA380
Device: Continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes — Continuous veno-venous hemodiafiltration (CVVHDF) with Oxiris®-AN69 membranes (control arm)
  Arms: CVVHDF with Oxiris®-AN69 membrane

SUMMARY:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. Intensive care unit (ICU) mortality in patients with septic shock and acute kidney injury (AKI) requiring continuous renal replacement therapy (CRRT) remains high and approximates 50-60%. Sepsis is the leading etiology for AKI and CRRT requirement in ICU patients.

In septic shock, the dysregulated host response to infectious pathogens leads to a cytokine storm with uncontrolled production and release of humoral pro-inflammatory mediators. These pro-inflammatory mediators and cytokines exert cellular toxicity and promote the development of organ dysfunction and increased mortality.

In addition to treating AKI, CRRT techniques can be employed for adsorption of inflammatory mediators extracorporally using specially developed adsorption membranes, hemoperfusion sorbent cartridges or columns. Several methods and devices, such as Oxiris®-AN69 membrane, CytoSorb® cytokine hemoadsorption and polymyxin B (Toraymyxin) endotoxin adsorption and plasmapheresis have been evaluated in small study series but to date the data on outcome benefits remains controversial.

HA380 (Jafron Biomedical Co , Ltd, Zhuhai, China) is a CE-labeled hemoadsorption cartridge developed to treat patients with septic shock. It contains hemo-compatible, porous polymeric beads that adsorp cytokines and mid-molecular weight toxins on their surface. The cytokines absorved using this cartridge are IL-1, IL-6, IL-8, IL-10 in addition to TNF-α8.

Therefore, this study aims to examine the potential effects of cytokine adsorption using HA380 in addition to hemodiafiltration with the Oxiris®-AN69 membrane on ICU- and 90-day mortality in patients with septic shock and AKI.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection and carries a risk for lethality, considerably exceeding that of a mere infection. Intensive care unit (ICU) mortality in patients with septic shock and acute kidney injury (AKI) requiring continuous renal replacement therapy (CRRT) remains high and approximates 50-60% despite recent technical advancements in patient care. Sepsis is the leading etiology for AKI and CRRT requirement in ICU patients and almost half of the critically ill patients with sepsis develop AKI.

In septic shock, the dysregulated host response to infectious pathogens leads to a cytokine storm with uncontrolled production and release of humoral pro-inflammatory mediators. These pro-inflammatory mediators and cytokines exert cellular toxicity and promote the development of organ dysfunction and increased mortality. Septic shock is defined according to the Sepsis-3 consensus criteria as sepsis with a vasopressor requirement to maintain a mean blood pressure (MAP) ≥65 mm Hg, despite adequate fluid resuscitation, and a serum lactate level >2 mmol/L.

In addition to treating AKI, CRRT techniques can be employed for adsorption of inflammatory mediators extracorporally using specially developed adsorption membranes, hemoperfusion sorbent cartridges or columns. The aim of these techniques is to decrease the early deleterious effects of the cytokine storm and high endotoxin levels during the first hours and days of treatment of septic shock to benefit the patient. Several methods and devices, such as Oxiris®-AN69 membrane, CytoSorb® cytokine hemoadsorption and polymyxin B (Toraymyxin) endotoxin adsorption and plasmapheresis have been evaluated in small study series or are under evaluation for improving patient outcomes in septic shock. However, to date the data on outcome benefits remains controversial. Previous study series have shown a decrease in cytokine levels, improved hemodynamics and diminished need for vasopressor in patients treated using these methods. However, mortality benefit remains unclear.

HA380 (Jafron Biomedical Co , Ltd, Zhuhai, China) is a CE-labeled hemoadsorption cartridge developed to treat patients with septic shock. It contains hemo-compatible, porous polymeric beads that adsorp cytokines and mid-molecular weight toxins on their surface. The cytokines absorved using this cartridge are IL-1, IL-6, IL-8, IL-10 in addition to TNF-α8.

Therefore, this study aims to examine the potential effects of cytokine adsorption using HA380 in addition to hemodiafiltration with the Oxiris®-AN69 membrane on ICU- and 90-day mortality in patients with septic shock. To study patients with the highest degree of morbidity the study will recruit only septic shock patients with a high vasopressor requirement before CRRT initiation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, admitted to the ICU
* Septic shock according to the Sepsis-3 criteria and a norepinephrine requirement ≥0.2µg/kg/min despite adequate fluid resuscitation
* Acute kidney injury at or after ICU admission and the treating physician considers that initiation of CRRT is likely within 48 hours.
* Informed consent from the patient or family members is received

Exclusion Criteria:

* Maintenance dialysis dependency or RRT during current hospital stay prior to ICU admission
* GFR less than 20ml/kg/1.73m2 prior to hospital admission (within 365 days)
* Neurosurgical patients
* Pregnant women
* Patient's lack of commitment to start RRT
* Chronic or acute clinical condition with a prognosis below 6 months
* History of heparin allergy or heparin induced thrombocytopenia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intensive care mortality | During ICU care, 1 year
  Intensive care mortality
90-day mortality | Within 90 days from ICU admission, 90 days
  90-day mortality
Days alive at day 90 without vasoactives, invasive mechanical ventilation and renal replacement therapy. | 90 days following ICU admission, 90 days
  Days alive at day 90 without vasoactives, invasive mechanical ventilation and renal replacement therapy.

SECONDARY OUTCOMES:
Vasopressor support at 24 hours, 48 hours and 72 hours following CVVHDF initiation | 24 hours, 48 hours and 72 hours following CVVHDF initiation
  Noradrenalin infusion rate (unit:µg/kg/min) at 24 hours, 48 hours and 72 hours following CVVHDF initiation
Fluid balance at 24 hours, 48 hours and 72 hours following CVVHDF initiation | 24 hours, 48 hours and 72 hours following CVVHDF initiation
  Cumulative fluid balance (unit: ml) at 24 hours, 48 hours and 72 hours following CVVHDF initiation
Cytokine levels at 24 hours, 48 hours and 72 hours following CVVHDF initiation | 24 hours, 48 hours and 72 hours following CVVHDF initiation
  Cytokine levels (unit: ng/l) at 24 hours, 48 hours and 72 hours following CVVHDF initiation
C-reactive protein levels at 24 hours, 48 hours and 72 hours following CVVHDF initiation | 24 hours, 48 hours and 72 hours following CVVHDF initiation
  C-reactive protein levels (unit: mg/l) at 24 hours, 48 hours and 72 hours following CVVHDF initiation
Procalcitonin levels at 24 hours, 48 hours and 72 hours following CVVHDF initiation | 24 hours, 48 hours and 72 hours following CVVHDF initiation
  Procalcitonin levels (unit: µg/l) at 24 hours, 48 hours and 72 hours following CVVHDF initiation
Renal recovery at 90-days following randomization | 90 days following randomization, 90 days
  Estimated glomerular filtration rate (unit: ml/min/1.73 m²) and dialysis dependency (yes/no) at 90-days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Mikko J Järvisalo, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No